CLINICAL TRIAL: NCT02104271
Title: Comparison Between Two Different Parameters of Argon Plasma Coagulation in the Treatment of Chronic Radiation Proctitis: Historical Control Trial.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Denise Peixoto Guimarães, MD, PhD, Barretos Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 662/2012
Record Dates: First submitted 2014-03-13; First posted 2014-04-04 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Radiation Injuries; Telangiectasis; Rectal Bleeding
Keywords: chronic radiation proctitis; argon plasma coagulation; rectal bleeding
MeSH Terms: conditions — Radiation Injuries; Telangiectasis; Gastrointestinal Hemorrhage | interventions — Argon Plasma Coagulation; Lasers, Gas; Historically Controlled Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Argon Plasma Coagulation (Experimental): Argon Plasma Coagulation (APC) treatment will be delivered using a "spray-painting" technique, with short applications at 40W power and argon gas flow of 1.2 L/min. The APC equipment consists of a high frequency electrosurgical generator combined with a source of argon gas (Argon + SS601MC 4 , WEM Electronic Equipment Ltda , Ribeirão Preto , Brazil ). A flexible catheter of 2.3 mm diameter ( WEM ) Teflon coated and with a hint of heat resistant ceramic is inserted through the working channel of the colonoscope and connected to the current generator and the gas source for APC implementation.
  Interventions: Procedure: Argon Plasma Coagulation
- Historical control (Active Comparator): Argon Plasma Coagulation (APC) treatment was delivered using a "spray-painting" technique, with short applications at 40-50W power and argon gas flow of 2.0 - 2.5 L/min. The APC equipment consists of a high frequency electrosurgical generator combined with a source of argon gas (Argon + SS601MC 4 , WEM Electronic Equipment Ltda , Ribeirão Preto , Brazil ). A flexible catheter of 2.3 mm diameter ( WEM ) Teflon coated and with a hint of heat resistant ceramic is inserted through the working channel of the colonoscope and connected to the current generator and the gas source for APC implementation.
  Interventions: Procedure: Historical control

INTERVENTIONS:
Procedure: Argon Plasma Coagulation — APC was performed during sigmoidoscopy exam. Bowel preparation begins on the eve of the exam associated with waste liquid diet without oral intake of 10mg of bisacodyl (5mg/dragee) at 14 o'clock and 18pm and 130ml of phosfoenema (16g of sodium phosphate monobasic monohydrate and 6g of sodium phosphate dibasic heptahydrate per 100ml) diluted in 100ml of orange juice or lemon to 19h. On the day of the exam is administered 130ml of phosfoenema rectally immediately before the exam.
  All patients were previously sedated with fentanyl (0.05mg/ml), midazolam (5mg/5ml) and propofol (10mg/ml) and have intravenous introduction of the flexible colonoscope to the transverse colon to the exchange of gases following the routine of the Department of Endoscopy, Cancer Hospital Barretos.
  Other Names: Argon gas
  Arms: Argon Plasma Coagulation
Procedure: Historical control — APC was performed during sigmoidoscopy exam. Bowel preparation begins on the eve of the exam associated with waste liquid diet without oral intake of 10mg of bisacodyl (5mg/dragee) at 14 o'clock and 18pm and 130ml of phosfoenema (16g of sodium phosphate monobasic monohydrate and 6g of sodium phosphate dibasic heptahydrate per 100ml) diluted in 100ml of orange juice or lemon to 19h. On the day of the exam is administered 130ml of phosfoenema rectally immediately before the exam.
  All patients were previously sedated with fentanyl (0.05mg/ml), midazolam (5mg/5ml) and propofol (10mg/ml) and have intravenous introduction of the flexible colonoscope to the transverse colon to the exchange of gases following the routine of the Department of Endoscopy, Cancer Hospital Barretos.
  Other Names: Argon gas
  Arms: Historical control

SUMMARY:
There is a wide variability of options for treatment of chronic radiation proctitis. However, studies are still limited, usually case reports from a single center and few are comparative studies between methods. Therefore, the choice of treatment is determined by availability and local expertise for each method. The variability of treatment options range from anti-inflammatory medical treatment, sucralfate, short chain fatty acids, antioxidants and hyperbaric oxygen to such endoscopic and surgical treatments. Surgery is usually the last therapeutic option due to the high morbidity and mortalityassociated. Various endoscopic treatment modalities have been reported. Formalin topic is effective in up to 48% of patients with chronic radiation proctitis.

The endoscopic treatment with argon plasma (APC) is low cost, easy to apply and transportation, safe and effective in the treatment of rectal bleeding in patients with chronic radiation proctitis. Currently, the APC is the preferred endoscopic modality.

Most studies on the use of APC in radiation proctitis showed benefit. The APC controls the mild to moderate rectal bleeding in 80% to 90% of cases and improves symptoms of urgency, diarrhea and tenesmus in 60% to 75% of cases.

DETAILED DESCRIPTION:
APC is usually applied with a power of 40-60W and 1.2-2.5 L/min of gas flow by using a electrosugical generator coupled with an argon delivery unit. However, high gas flow have been associated to high rates of complication such as rectal stenosis and deep rectal ulcer.

In this context, the present study aims to compare the effectiveness and safety between two different paramenters of argon plasma coagulation (40-50W and 2.0 L/min of gas flow vs 40W and 1.2 L/min of gas flow) in the treatment of patients with symptomatic chronic radiation proctitis.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* endoscopic diagnosis of chronic radiation proctitis
* previous pelvic radiotherapy
* presence of colonic or rectal telangiectasias
* patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* other causes of rectal bleeding besides chronic radiation proctitis diagnosed by complete colonoscopy , such as colorectal cancer , inflammatory bowel disease and polyps larger than 1 cm
* use of oral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Rectal bleeding rates | Up to four weeks after the administration of the first dose of APC and every four weeks after that up to 24 weeks
  The proportion of patients with Complete Response at Week 4, 8, 12, 16, 20 and 24 defined as absence of bleeding.
Occurrence of rectal ulcers | Up to four weeks after the administration of the first dose of APC and every four weeks after that up to 24 weeks.
  Presence of detectable rectal ulcers (>10mm size or deep ulcers) on endoscopy.

SECONDARY OUTCOMES:
Recurrence of rectal bleeding | 6 and 12 months after the administration of the last dose of APC
  Abscence or recurrence of rectal bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil